CLINICAL TRIAL: NCT05730673
Title: A Phase II Study of Leronlimab (PRO 140) in Combination With Regorafenib in Patients With CCR5+, Microsatellite Stable (MSS), Metastatic Colorectal Cancer (mCRC)
Brief Title: Leronlimab in Combination With Regorafenib in Patients With CCR5+, Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: CytoDyn, Inc. (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD08_mCRC
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: CCR5; Microsatellite Stable; Metastatic; Colorectal Cancer
Keywords: Metastatic; Colorectal Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Leronlimab in combinatiob with Regorafenib (Experimental): Leronlimab (PRO 140) will be administered subcutaneously at a weekly dose of 700 mg in combination with staring dose of 80 mg Regorafenib at first week of the Cycle 1, followed by escalation of Regorafenib dose to 120 mg and 160 mg in second and third weeks of Cycle 1, respectively. No Regorafenib will be administered during the fourth week.
  Interventions: Drug: 700mg leronlimab weekly dose; Drug: 80mg Regorafenib at week 1; Drug: 120mg Regorafenib at week2; Drug: 160 mg Regorafenib at week 3

INTERVENTIONS:
Drug: 700mg leronlimab weekly dose — leronlimab is a humanized IgG4,κ monoclonal antibody (mAb) to the chemokine receptor CCR5
Drug: 80mg Regorafenib at week 1 — Regorafenib is a small-molecule multiple kinase inhibitor
Drug: 120mg Regorafenib at week2 — Regorafenib is a small-molecule multiple kinase inhibitor
Drug: 160 mg Regorafenib at week 3 — Regorafenib is a small-molecule multiple kinase inhibitor

SUMMARY:
This is aPhase II Study of Leronlimab (PRO 140) in combination with Regorafenib in Patients with CCR5+, Microsatellite Stable (MSS), Metastatic Colorectal Cancer (mCRC)

DETAILED DESCRIPTION:
This ia a phase II, single arm study with 30 patients in order to test the hypothesis that the combination of Leronlimab (PRO 140) SC and oral Regorafenib will increase PFS in patients with CCR5 + MSS mCRC.

Leronlimab will be administered subcutaneously at a weekly dose of 700 mg in combination with staring dose of 80 mg Regorafenib at first week of the Cycle 1, followed by escalation of Regorafenib dose to 120 mg and 160 mg in second and third weeks of Cycle 1, respectively. No Regorafenib will be administered during the fourth week.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient age ≥ 18 years with a history of treated colorectal cancer with unresectable metastases of the primary colorectal cancer to the other organs.
2. Demonstrate CCR5 + by IHC (>10% membranous staining completed at the reference laboratory of Dr. Hallgeir Rui at Medical College of Wisconsin).

   Note: This test will be done as part of the pre-screening period. It will be performed in archival metastatic tissue.
3. Histologically confirmed for microsatellite stable MSS colorectal cancer by Immunohistochemistry (IHC) or Next-generation sequencing (NGS)
4. Metastatic colorectal cancer (CRC) who have been previously treated with fluoropyrimidine-, oxaliplatin- and irinotecan-based chemotherapy, VEGF antibody, and, if RAS wild-type, an anti-EGFR therapy Note: Prior Regorafenib therapy is not allowed.
5. Have measurable disease per RECIST 1.1
6. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Expected survival of at least three months
9. No chemotherapy treatment within the last four weeks or less than wash out period of the chemotherapy agents, whichever is shorter
10. Patients must have adequate organ and bone marrow function within 28 days prior to registration, as defined below:

    * Leukocytes ≥ 3,000/mcL;
    * Absolute neutrophil count ≥ 1,500/mcL;
    * Platelet count > 75,000/mm^3
    * Total bilirubin: within normal institutional limits;
    * AST(SGOT) &ALT(SPGT) ≤ 2.5 X institutional upper limit of normal (ULN) (applicable to all patients, irrespective of liver disease or metastasis); and
    * Creatinine: within normal institutional limits.
11. Clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator.
12. Both male and female patients and their partners of childbearing potential must agree to use two medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], or one of the following methods of birth control (intrauterine devices, tubal sterilization or vasectomy) or must practice complete abstinence from intercourse of reproductive potential from study entry to 6 months after the last day of treatment (excluding women who are not of childbearing potential and men who have been sterilized).
13. Females of child-bearing potential (FOCBP) must have a negative serum pregnancy test at Screening Visit and negative urine pregnancy test prior to receiving the first dose of study drug; and
14. Male participants must agree to use contraception and refrain from donating sperm for at least 120 days after the last dose of study intervention.
15. Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study.

Exclusion Criteria:

1. Inability to understand the aims of the study and/or protocol procedures
2. Hypersensitivity towards Regorafenib or Leronlimab (PRO 140).
3. History of severe allergic, anaphylactic, or other hypersensitivity reactions to humanized monoclonal antibodies
4. Any other concurrent antineoplastic treatment including irradiation (local radiation of single non-target lesions for palliation only allowed)
5. Any condition requiring continuous systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 2 weeks prior to first dose of study treatment. Inhaled or topical steroids and physiological replacement doses of up to 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
6. Clinically significant active coronary heart disease and cardiovascular insufficiency with hypotension (systolic blood pressure <100 mmHg) per PI discretion.
7. Cardiac arrhythmias requiring anti-arrhythmic therapy; Note: pace makers, beta blockers, or digoxin are permitted
8. Any GI or Respiratory system disorders that per PI discretion can interfere with the study treatment or jeopardize the patient's health.
9. Prior allogeneic bone marrow transplantation
10. Administration of a live, attenuated vaccine within four weeks prior to start of maintenance treatment or anticipation that such a live attenuated vaccine will be required during the remainder of the study Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
11. Positive test for human immunodeficiency virus (HIV) or HIV infection
12. Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test) or hepatitis C. Note: Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible.
13. Active or latent tuberculosis
14. Clinically active brain metastases, defined as untreated symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms.
15. Patient who have an active infection requiring systemic therapy.
16. Patient who are taking strong CYP3A4 inducers (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, and St. John's Wort) or strong CYP3A4 inhibitors (e.g. clarithromycin, grapefruit juice, itraconazole, ketoconazole, nefazodone, posaconazole, telithromycin, and voriconazole)
17. Are pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the Screening Visit through 120 days after the last dose of study intervention.
18. Have undergone major surgery and have not recovered adequately from any toxicity and/or complications from the intervention before starting study intervention.
19. Have a seizure disorder requiring ongoing antiseizure therapy or with any condition that, in the judgment of the investigator, is likely to increase the risk of seizure (e.g., CNS malignancy.)
20. Have received prior therapy with Leronlimab or any other CCR5 antagonist (e.g., maraviroc).
21. Have received prior therapy with regrafenib.
22. Have been treated with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX 40, CD137).
23. Patient who received prior radiotherapy (not to target lesions) within 3 weeks of start of study intervention.
24. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 28 days prior to enrollment;
25. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-20 (Estimated); Primary Completion 2023-05-27 (Estimated); Study Completion 2023-08-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR, defined as Complete Response (CR) + Partial Response (PR)) in subjects with CCR5+ mCRC treated with Leronlimab (PRO 140) and Regorafenib. | Four weeks

SECONDARY OUTCOMES:
The number, frequency, and severity of adverse events (AEs) collected from the time of first treatment until 12 weeks after study treatment completion to evaluate safety of Leronlimab (PRO 140) and Regorafenib in subjects with CCR5+ mCRC. | Four weeks
Progression free survival (PFS) defined as time in months from the date of first study treatment to the date of disease progression or death from any cause, whichever comes first. | Four weeks
Overall survival defined as time in months from the date of first study treatment to the date of death; | Four weeks
Time to new metastases (TTNM) | Four weeks
The change from baseline in circulating tumor cells (CTC) in the peripheral blood. | Four weeks

OTHER OUTCOMES:
Measure serum level of CCL2, CCL3, CCL4 and CCL5 and correlate with therapeutic benefit (PFS) in patient with mCRC. | Four weeks